CLINICAL TRIAL: NCT00796185
Title: Comparison of Steady-state Pharmacokinetics of Paliperidone After Extended-release OROS� Paliperidone 15 mg and Immediate-release Oral Risperidone 8 mg b.i.d. in Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: As Study of the Pharmacokinetics of Paliperidone Extended-release and Risperidone Immediate-release Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004270
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Mood Disorders; Antipsychotic drugs; Paliperidone ER
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mood Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone ER

SUMMARY:
The purpose of this study is to compare the steady-state pharmacokinetics of paliperidone after oral administration of 15 mg extended-release (ER) OROS paliperidone once daily with the steady-state pharmacokinetics of paliperidone after oral administration of 8 mg immediate-release (IR) risperidone twice daily; and to explore the dose-proportionality of 9 mg and 15 mg ER OROS paliperidone. Other objectives are to 1) document the disposition of the enantiomers of paliperidone; 2) explore the relationship between genotype (CYP2D6, CYP3A4, CYP3A5, UGT1A1, and UGT1A6) and pharmacokinetic parameters; and 3) assess safety and tolerability.

DETAILED DESCRIPTION:
This is an open-label, multiple-dose, parallel-group study in patients with schizophrenia or schizoaffective disorder. The study consists of a screening period (2 weeks maximum); a 1-week run-in or washout (Days 1 to 7) during which patients taking risperidone prestudy and randomly assigned to paliperidone treatment will receive replacement antipsychotic therapy, and other patients continue to take their prestudy antipsychotic medication; a 14-day open-label treatment period (Days 8 to 21); and a 5-day follow-up period. On Day 1 of the washout period, eligible patients will be randomized to receive ER OROS paliperidone (PAL) or risperidone (RIS). All patients will receive their first dose of study medication on Day 8 after randomization as follows: Patients randomized to PAL will receive 9 mg of ER OROS paliperidone daily from Day 8 to Day 14, followed by 15 mg of ER OROS paliperidone q.d. from Day 15 to Day 21. Patients randomized to RIS will receive dose-escalation up to 7 mg risperidone twice daily (b.i.d.) from Day 8 to Day 14, followed by 8 mg risperidone b.i.d. from Day 15 to Day 21. The study medication on Days 14 and 21 in the PAL group and on Day 21 in the RIS group will be administered after completion of a standardized high fat, high caloric breakfast. Patients will be confined to the testing facility from the morning of Day 8 (or earlier at the discretion of the investigator) until completion of the study procedures on Day 23. On all other assessment days, patients will return to the testing facility and remain there for the duration of the assessments.The highest dose of paliperidone currently being studied is 12 mg given as 6 tablets of 2 mg ER OROS paliperidone. In the currently proposed study, data on the safety and tolerability of the 15-mg dose will be monitored and collected. Paliperidone ER oral administration of 9 mg q.d. on Day 8 to 14, and 15 mg daily on Day 15 to 21; oral administration of escalating doses up to 7 mg risperidone twice daily (b.i.d.) between Days 8 and 14, inclusive, and 8 mg risperidone b.i.d. on Day 15 to 21

ELIGIBILITY:
Inclusion Criteria:

* Currently treated with a dose of at least 6 mg of risperidone daily or the equivalent of any other antipsychotic medication or a combination thereof (an equivalence table will be provided to the sites)
* Has a DSM-IV diagnosis of schizophrenia (295.10, 295.20, 295.30, 295.60, 295.90) or schizoaffective disorder
* Healthy on the basis of a prestudy physical exam, medical history, ECG, and laboratory results of blood biochemistry, hematology, and urinalysis performed within 2 weeks of randomization. If the results of the biochemistry or hematology tests or the urinalysis are not within the laboratory's reference ranges the patient can be included only if the investigator judges that the deviations are not clinically significant. For liver function tests (alanine transaminase, aspartate transaminase, and bilirubin), the values must be contained within 2 times the upper limits of the normal laboratory reference ranges and for renal function tests, the values must be within the normal laboratory reference ranges
* Women must be postmenopausal for at least 1 year, surgically sterile, or practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization and at the discretion of the investigator, total abstinence) before entry and throughout the study, as well as have a negative serum pregnancy test at screening. To ensure continued eligibility, women must have a negative urine test at baseline
* Body weight as defined by body mass index (weight [kg]/height (m)²) within a range of 15.0 to 35.0 kg/m², inclusive
* Willingness to spend 15 days as an in-patient during the treatment period
* Normotensive at screening, with supine (5 minutes) blood pressure between the range of 100 to 140 mmHg systolic, inclusive, and 60 to 90 mmHg diastolic, inclusive.

Exclusion Criteria:

* Involuntarily committed in-patients
* Has a DSM-IV diagnosis of substance dependence within 3 months before screening evaluation. Nicotine and caffeine dependence and history of recreational use of marijuana are not exclusionary
* At screening, has a decrease of > = 20 mmHg systolic blood pressure or a decrease of > =10 mmHg decrease in diastolic blood pressure 2 minutes after standing, or experience symptoms of lightheadedness, dizziness, or fainting upon standing
* orthostatic hypotension
* Tests positive for the urine drug screen at screening
* Had an acute exacerbation of psychotic symptoms within the last 3 months before screen
* Relevant history or current presence of any cardiovascular, respiratory, central nervous system, neuropsychiatric (including seizures), renal, hepatic, endocrine, or immunologic diseases
* Has a DSM-IV Axis I diagnosis other than schizophrenia or schizoaffective disorder
* Suicidal or homicidal ideation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2003-08; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
To compare the steady-state pharmacokinetics of paliperidone after administration of ER OROS paliperidone at 15 mg orally and IR risperidone at 8 mg orally, twice daily; to explore the dose-proportionality of 9 mg and 15 mg paliperidone ER

SECONDARY OUTCOMES:
To document the disposition of the enantiomers of paliperidone, to explore the relationship between genotypes (CYP2D6, CYP3A4, CYP3A5, UGT1A1, and UGT1A6) and pharmacokinetic parameters, and to assess safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: As study of the pharmacokinetics of paliperidone extended-release and risperidone immediate-release formulations — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=575&filename=CR004270_CSR.pdf